CLINICAL TRIAL: NCT03945721
Title: A Phase I Study of Niraparib Administered Concurrently With Postoperative RT in Triple Negative Breast Cancer Patients (UNITY)
Brief Title: A Phase I Study of Niraparib Administered Concurrently With Postoperative RT in Triple Negative Breast Cancer Patients
Acronym: UNITY
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Principal Investigator, Steven J Isakoff, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-055
Record Dates: First submitted 2019-04-29; First posted 2019-05-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer; Residual Disease
Keywords: Breast Cancer; Triple Negative; Locally Advanced
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm, Residual; Breast Neoplasms | interventions — niraparib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental): * Niraparib will be administered orally on a daily basis
  * Radiation Therapy will be administered concurrently with Niraparib
  Interventions: Drug: Niraparib; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Niraparib — Niraparib is a type of drug called a "PARP inhibitor", which blocks DNA (the genetic material of cells) damage from being repaired or may prevent damage from occurring in the first place. In cancer treatment, inhibiting PARP may help kill cancer cells by not allowing the cancer cells to repair its DNA damage or prevent DNA damage from occurring.
Radiation: Radiation Therapy — radiation therapy

SUMMARY:
This research study involves Niraparib as a possible treatment for triple negative breast cancer.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved niraparib for this specific disease but it has been approved for other uses.

Niraparib is a type of drug called a "PARP inhibitor", which blocks DNA (the genetic material of cells) damage from being repaired or may prevent damage from occurring in the first place. In cancer treatment, inhibiting PARP may help kill cancer cells by not allowing the cancer cells to repair its DNA damage or prevent DNA damage from occurring.

This trial is studying people who have triple negative breast cancer because this cancer type is shown to have DNA repair mechanisms that may benefit from combined PARP inhibitor and radiation, and may help prevent recurrence of cancers in the chest wall and lymph nodes of the affected side.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females, ≥ 18 years of age.
* Non-metastatic, histologically or cytologically-confirmed TNBC (defined as ER <1%, PR <1%, her-2-neu 0-1+ by IHC or FISH-negative or as per MD discretion).
* Definitive surgical treatment with breast-conserving surgery or mastectomy and axillary lymph node evaluation.
* Plans for receipt of postoperative radiation therapy to the breast/chest wall +/- regional nodes
* Residual invasive disease after NAC (any size), or at least 1.0 cm in patients who do not receive NAC and undergo surgery first.
* ECOG Performance status ≤ 1.
* Willingness to discontinue any cytotoxic chemotherapeutic agents, immunotherapy and biologic therapy at least 2 weeks prior to the start of RT.
* Adequate organ function (assessed within 30 days prior to initiation of protocol treatment, unless otherwise indicated) as follows:

  * Hematology
  * Absolute Neutrophil Count (ANC) ≥1500/mm3
  * Platelet Count ≥100,000/mm3
  * Hemoglobin ≥9.0 g/dL
  * Renal Function
  * Creatinine Serum ≤ 1.5 mg/dL or
  * Creatinine Clearance ≥ 45 mL/mina
  * Hepatic Function
  * Bilirubin ≤ 1.5 mg/dL
  * Aspartate Aminotransferase (AST) ≤ 2.5 x ULNb
  * Alanine Aminotransferase (ALT) ≤ 2.5 x ULN
  * ULN = upper normal limit of institution's normal range
  * If calculated creatinine clearance is < 45mL/min, a 24-hour urine collection for creatinine clearance may be performed
  * Subjects with documented Gilbert's disease may have bilirubin up to 2.5 mg/dL
* Female participants have a negative urine or serum pregnancy test within 7 days prior to study treatment if a woman has child-bearing potential, and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of non-childbearing potential.
* Non-childbearing potential is defined as follows (by other than medical reasons):

  --≥45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. See Section 5.6.4.5 for a list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Male participant agrees to use an adequate method of contraception (see Section 5.6.4.5) for a list of acceptable birth control methods) starting with the first dose of study treatment through 90 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Participant must agree not to breastfeed during the study or for 30 days after the last dose of study treatment.
* Participant receiving corticosteroids may continue as long as their dose is stable for at least 4 weeks prior to initiating protocol therapy.
* Participant must agree not to donate blood during the study or for 90 days after the last dose of study treatment.
* Ability to swallow (whole) and retain oral medications.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Dose Cohort 2 only:

  * Actual body weight ≥77kg AND
  * Platelet count ≥150,000 µL

Exclusion Criteria:

* Gross residual tumor or positive margins after surgery that is un-excised (excluding positive margins at the chest wall or skin where no additional breast tissue can be removed).
* pT1aN0 or pT1bN0 (primary tumor size <1.0 cm) triple negative breast cancer patients who do undergo neoadjuvant chemotherapy and receive surgery followed by +/- adjuvant chemotherapy.
* Receipt of PARP inhibitor at any time prior to study enrollment.
* Pregnant or expecting to conceive within the projected duration of the trial, starting with screening visit through 180 days after the last dose of trial treatment.
* Prior history of radiation therapy to the ipsilateral breast and/or regional nodes is not allowed (prior RT to other sites that was completed ≥ 1 week prior to Day 1 of protocol therapy, or if prior RT encompassed >20% of the bone marrow it was completed ≥ 2 weeks prior to Day 1 of protocol therapy, is permitted).
* Major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to niraparib, or its components or excipients.
* Concomitant anti-neoplastic treatment is not allowed during protocol treatment and should be completed at least 2 weeks prior to commencement of protocol treatment, with resolution of associated acute toxicities. Bisphosphonates are permitted without restriction even during protocol treatment.
* Significant comorbidity: Patients with clinically significant and uncontrolled major disease or disorder that could exacerbate potential toxicities, confound safety assessments, require excluded therapy for management, or limit study compliance.
* Treatment with investigational therapy within ≤ 4 weeks, or within a time interval less than at least five half-lives of the investigational agent, whichever is shorter, prior to initiating protocol therapy. Patients may not be simultaneously enrolled in any interventional clinical trial.
* Unresolved toxicity from other agents. Patients with unresolved CTCAE v5 Grade 2 or greater toxicity, with the exception of alopecia and anemia, from prior administration of another investigational drug and/or anti-cancer treatment are not eligible.
* Known grade 3 or 4 anemia, neutropenia, or thrombocytopenia that persisted > 4 weeks and was related to the most recent chemotherapy treatment.
* Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
* Participant must not have received colony-stimulating factors (e.g. granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior to initiating protocol therapy.
* Prior malignancy within 5 years of study enrollment.
* Scleroderma and systemic lupus erythematosis.
* Known p53 germline mutations.
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Known symptomatic brain or leptomeningeal metastases.
* Dose Cohort 2 only:

  * Actual body weight < 77kg OR
  * Platelet count < 150,000 µL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 10 weeks
  The proportion of subjects tolerating each maximum dose level. The trial will be monitored using a 3+3 dose escalation method.

SECONDARY OUTCOMES:
Locoregional Relapse | 2 years
  The incidence of recurrence of breast cancer in the ipsilateral chest wall or regional lymph nodes will be captured
Distant Relapse | 2 years
  The incidence of recurrence of breast cancer in regions outside of the ipsilateral chest wall or regional lymph nodes will be captured
Treatment related adverse events | 2 Years
  Adverse events will be assessed using common terminology criteria for adverse events (CTCAE) v5.
Breast cosmesis | 2 years
  Breast cosmesis will be assessed using the Radiation Therapy Oncology Group (ROTG) cosmesis assessment criteria. Brest cosmesis will be reported as the number of participants reporting excellent/good or fair/poor cosmetic results.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Ho, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute/Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation